CLINICAL TRIAL: NCT04463264
Title: Efficacy and Safety Study of Nitazoxanide (NTX) in the Treatment of Patients With SARS-CoC-2 Virus Infection (COVID-19). A Pilot, Randomized, Simple Blind, Placebo-controlled, Parallel-group Study
Brief Title: Efficacy and Safety Study of Nitazoxanide (NTX) in the Treatment of Patients With SARS-CoV-2 Virus Infection (COVID-19)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Roemmers S.A.I.C.F. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTZ-COVID ARG1
Record Dates: First submitted 2020-06-26; First posted 2020-07-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Nitazoxanide; Coronavirus Infections; RNA Virus Infections; Respiratory Tract Infections; Virus Diseases; Respiratory Tract Diseases; Antiparasitic Agents
MeSH Terms: conditions — COVID-19; Coronavirus Infections; RNA Virus Infections; Respiratory Tract Infections; Virus Diseases; Respiratory Tract Diseases | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Randomized. Nitazoxanide : Placebo (2:1), parallel-group study
Who Masked: Participant
Masking Description: Simple blind design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTX active treatment (Experimental): Intervention: NTX (500 mg every 6 hours for 14 days) orally with food (P.O.).
  Interventions: Drug: Nitazoxanide
- Intervention: placebo (Placebo Comparator): Placebo (1 tablet every 6 hours for 14 days) orally with food (P.O.).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — NTX (500 mg every 6 hours for 14 days) orally with food (P.O.).
  Arms: NTX active treatment
Drug: Placebo — Placebo (1 tablet every 6 hours for 14 days) orally with food (P.O.).
  Arms: Intervention: placebo

SUMMARY:
Evaluation of the efficacy and safety of NTX in adult patients (≥18 years and <60 years), with SARS-CoV-2 infection with mild symptoms of COVID-19, compared to a placebo control arm. 135 patients will be randomized to either Nitazoxanide (n=90) or placebo (n=45) (2:1). Simple blind design. Primary endpoint: eradication of virus from patients' respiratory tract secretions by the 7th day of treatment.

DETAILED DESCRIPTION:
The rapid spread of COVID-19 has overwhelmed the capabilities of the Public Health System in major nations due to the large number of critically ill patients and patients seriously affected requiring intensive care.

Reducing the viral load, along with other epidemiological measures, including social isolation and quarantine, may in the long run significantly reduce the R0 (Basic Reproductive Rhythm) of infection.

To date, in our country there are no specific antiviral treatments approved by the regulatory authorities for COVID-19, and no vaccines so far exist. Symptomatic and supportive treatment has been the main intervention for patients with moderate to severe infection.

The lack of a drug with a demonstrated solid antiviral efficacy warrants the need to explore new therapeutic options against SARS-CoV-2 / COVID-19.

Nitazoxanide is a widely used thiazolide, approved by the FDA and ANMAT (Argentine drug regulatory authority) as an antiprotozoal, with a very good safety record for a variety of indications. NTX was shown to have extensive antiviral activity against, inter alia, animal and human coronaviruses. Indeed, it exhibits in vitro activity against MERS-CoV and other coronaviruses, including SARS-CoV-2, where it inhibits the expression of viral protein N. Another proposed antiviral mechanism for Nitazoxanide involves PKR and eIF2α phosphorylation and the depletion of ATP-sensitive intracellular calcium deposits in infected cells, thereby inducing chronic sub-lethal stress of the endoplasmic reticulum and impairing the glycosylation of the structural protein.

Exposure in clinical trials included a specific experience on patients with uncomplicated influenza-like illness, where the drug helped reduce the mean time for symptom relief.

The objective of this study is to evaluate the efficacy and safety of NTX (1,000mg/3 times per day plus standard treatment for 14 days in male and female patients (≥ 18 years and <60 years) with COVID-19 infection, with mild symptoms, as compared to a control group treated with placebo. The proposed study dose regime of Nitazoxanide 1,000 mg/3 times per day (every 8 hours) for 14 days may be modified if patients experience considerable GI adverse effects. In these cases, the dose may be lowered to one (1) 500 mg tablet every 6 hours (2,000 mg /day). Nitazoxanide has been also administered in other studies up to 4 g daily without significant adverse effects or changes in ECG or other laboratory values.

The proposed treatment regimen is expected to reduce disease severity by earlier eradication of viral load in NTX-treated patients when compared to placebo-treated patients, thus preventing the dysregulation of the innate immune system caused by the viral infection and modifying the high mortality in older/vulnerable populations. Early virus negativization or viral load reduction can potentially reduce the severity of the symptoms, eventually preventing a liable collapse of the Health Care System and ensuring a more controlled response to the disease.

Because of its known antiviral and safety profiles, and the fact that it can be orally administered to both adults and children, as well as its rapid availability and affordability, Nitazoxanide appears as an interesting alternative for such a situation.

Statistical analysis: 1-tailed statistical test, with a 25% α value (or type I error) (p value <0.025) and a power (type II error, or β value) of 0.20 (power of 80%) for superiority of the intervention arm over the control arm. All statistical analyzes will be carried out using STATA, version 14.0.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients (≥ 18 years and <60 years).
* Signature of informed consent.
* Patients with a positive test for SARS-CoV-2 and mild symptoms of COVID-19 (without severity criteria as detailed by the Ministry of Health of Argentina - MSN)

Exclusion Criteria:

* Patients under 18 years of age and over 60 years of age.
* Breastfeeding or pregnant women (with positive pregnancy blood test in women of childbearing age).
* Patients with mild pneumonia in the presence of risk factors or moderate or severe pneumonia (based on the severity criteria set by the Ministry of Health of Argentina), or patients who require mechanical ventilation at screening.
* Patients in whom NTX and/or lactose is contraindicated.
* Any other contraindication based on the judgment of the treating physician.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-26 (Estimated)

PRIMARY OUTCOMES:
Eradication of SARS COV-2 from patients' respiratory tract secretions by treatment day 7th. | 7 day
  Erradication will be considered a reduction of the viral load on day 7 greater than 35% with respect to placebo. Extraction of genomic material will be performed using a QIAgen mini kit (QIAmp viral RNA) validated by the CDC (United States Center for Disease Control and Prevention (https://www.fda.gov/media/134922/download) (CDC-006-00019) Viral load will be quantified with the following detection kits: Commercial Kit: PCR-EUA-CDC-nCoV-IFU. Commercial KIT SENTINEL - STAT-NAT Covid 19B (Berlín).
  Rational: In mild cases of COVID-19, 50% of the patients eradicated the virus within a period of 3 weeks, 25% eradicated the virus before the 13th day, 75% during the first month and the rest were " late eradicators." This latter subgroup of patients has been associated with severe cases of COVID-19 disease.

SECONDARY OUTCOMES:
Comparative decrease of the viral load | 3 - 35 days
  Consequently, in mild cases, viral eradication will likely occur more frequently during the first to second week of COVID-19 disease; less than 15% could eradicate the virus during the first week of symptom onset. From an epidemiological point of view, increasing the viral eradication rate from less than 15% to more than 35% during the first two weeks of treatment would be clinically relevant.(seven), 14 (fourteen) and 35 (thirty-five) after starting treatment compared to the baseline measurement.
Clinical improvement | 1 - 35 days
  Clinical improvement according to the WHO COVID-19 ordinal scale. Minimun 0 (zero), (best), maximum 8 (eight) (worst)
Pneumonia patients meeting severity criteria. | 1 - 35 days
  Percentage of pneumonia patients meeting severity criteria.
Number of days with fever | 1 - 35 days
  Number of days with fever (axillary temperature higher than 37.5°C).

OTHER OUTCOMES:
Patients requiring mechanical ventilation | 1 - 35 days
  Percentage of patients requiring mechanical ventilation through orotracheal intubation (OT) and/or ICU hospitalization.
Mortality rate. | 1- 35 days
  Mortality rate.
Lymphocyte recovery | 7 day
  Lymphocyte recovery (absolute lymphocyte count > 1000 / mm3).
ICU hospitalization. | 1 - 35 days
  Days of ICU hospitalization.
Oxygen saturation | 1 - 35 days
  Oxygen saturation (SpO2) > 92% (at ambient FiO2).
Days of hospitalization | 1 - 35 days
  Days of hospitalization
Respiratory rate | 1 - 35 days
  Respiratory rate per minute (in afebrile state conditions).

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Silva, MD, Principal Investigator — Austral University, Argentina
Locations (1):
- Hospital Universitario Austral, Presidente Derqui, Buenos Aires, Argentina, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashiru O, Howe JD, Butters TD. Nitazoxanide, an antiviral thiazolide, depletes ATP-sensitive intracellular Ca(2+) stores. Virology. 2014 Aug;462-463:135-48. doi: 10.1016/j.virol.2014.05.015. Epub 2014 Jun 25. PMID 24971706
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Chen J, Lau YF, Lamirande EW, Paddock CD, Bartlett JH, Zaki SR, Subbarao K. Cellular immune responses to severe acute respiratory syndrome coronavirus (SARS-CoV) infection in senescent BALB/c mice: CD4+ T cells are important in control of SARS-CoV infection. J Virol. 2010 Feb;84(3):1289-301. doi: 10.1128/JVI.01281-09. Epub 2009 Nov 11. PMID 19906920
- [Background] Chang D, Mo G, Yuan X, Tao Y, Peng X, Wang FS, Xie L, Sharma L, Dela Cruz CS, Qin E. Time Kinetics of Viral Clearance and Resolution of Symptoms in Novel Coronavirus Infection. Am J Respir Crit Care Med. 2020 May 1;201(9):1150-1152. doi: 10.1164/rccm.202003-0524LE. No abstract available. PMID 32200654
- [Background] Frieman M, Baric R. Mechanisms of severe acute respiratory syndrome pathogenesis and innate immunomodulation. Microbiol Mol Biol Rev. 2008 Dec;72(4):672-85, Table of Contents. doi: 10.1128/MMBR.00015-08. PMID 19052324
- [Background] Haffizulla J, Hartman A, Hoppers M, Resnick H, Samudrala S, Ginocchio C, Bardin M, Rossignol JF; US Nitazoxanide Influenza Clinical Study Group. Effect of nitazoxanide in adults and adolescents with acute uncomplicated influenza: a double-blind, randomised, placebo-controlled, phase 2b/3 trial. Lancet Infect Dis. 2014 Jul;14(7):609-18. doi: 10.1016/S1473-3099(14)70717-0. Epub 2014 May 19. PMID 24852376
- [Background] Jasenosky LD, Cadena C, Mire CE, Borisevich V, Haridas V, Ranjbar S, Nambu A, Bavari S, Soloveva V, Sadukhan S, Cassell GH, Geisbert TW, Hur S, Goldfeld AE. The FDA-Approved Oral Drug Nitazoxanide Amplifies Host Antiviral Responses and Inhibits Ebola Virus. iScience. 2019 Sep 27;19:1279-1290. doi: 10.1016/j.isci.2019.07.003. Epub 2019 Aug 8. PMID 31402258
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029